CLINICAL TRIAL: NCT03761654
Title: Detection of Myocardial Dysfunction in Non-severe Subarachnoid Hemorrhage (WFNS 1-2) Using Speckle-tracking Echocardiography (STRAIN)
Acronym: SAH-STRAIN
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2018/51
Record Dates: First submitted 2018-11-29; First posted 2018-12-03 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Subarachnoid Hemorrhage (SAH); Left Ventricular Dysfunction; Stress Cardiomyopathy
Keywords: Subarachnoid Hemorrhage (SAH); Left Ventricular Dysfunction; Intensive Care Unit; Speckle-tracking; STRAIN
MeSH Terms: conditions — Subarachnoid Hemorrhage; Ventricular Dysfunction, Left; Takotsubo Cardiomyopathy; Sprains and Strains

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with a "non-severe" subarachnoid hemorrhage
  Interventions: Diagnostic Test: Global Longitudinal Strain measure

INTERVENTIONS:
Diagnostic Test: Global Longitudinal Strain measure — Global Longitudinal Strain measure on day 1 of hospitalization

SUMMARY:
Subarachnoid hemorrhage (SAH) can cause transient myocardial dysfunction. Recently, it have been reported that myocardial dysfunctions that occur in SAH are associated with poor outcomes. It therefore appears essential to detect theses dysfunctions with the higher sensitivity as possible. Strain measurement using speckle-tracking echocardiography may detect myocardial dysfunction with great sensitivity. The main objective of this study is to assess the prevalence of myocardial dysfunction in "non-severe" SAH (defined by a WFNS grade 1 or 2), using speckle-tracking echocardiography. This study also aims to analyse Strain measurement with classical echocardiography and serum markers (troponin, BNP) of cardiac dysfunction.

DETAILED DESCRIPTION:
Cardiac complication, occurring in the early phase of SAH has been well described. It seems that the pathophysiological mechanism involves vegetative hyperactivity due to the acute cerebral injury. It has been shown that stress cardiomyopathy is associated with delayed cerebral ischemia (DCI) and poor outcomes. Manifestations of stress cardiomyopathy are changes in electrocardiogram, release of cardiac biomarkers such as troponin and BNP, and echography evidence of impaired left ventricle ejection fraction with the use of Simpson technique and regional wall motion abnormalities. These two techniques bear intra-observer variability. A new method is available to assess left ventricular contractility at the bedside. Two-dimensional speckle-tracking images with echocardiography allows one to track a natural myocardial marker within the myocardium by standard transthoracic echocardiography. It provides unique insights into myocardial function such as tissue deformations and strain rate, which is the rate of deformation. This method is more sensitive than classical echographic left ventricular ejection fraction evaluation and bears very low interobserver variability. The Global Longitudinal Strain (GLS) is the most studied parameter.

Early detection of cardiac dysfunction in SAH followed by appropriate monitoring and management may improve outcome in SAH. This is a prospective, observational and mono-center study.

Patients with "non-severe" SAH will benefit from an echocardiography where Left Ventricular Ejection Fraction (LVEF) and GLS will be assessed on day 1, 3 and 7 following the acute injury.

ELIGIBILITY:
Inclusion Criteria:

* patient older than 18 years
* hospitalized in neuro-intensive care unit with a "non-severe" subarachnoid hemorrhage (WFNS 1 or 2)

Exclusion Criteria:

* low echogenicity
* history of cardiac malformation or cardiac surgery
* severe valvular heart disease
* dilated cardiomyopathy
* acute coronary syndrome
* permanent arrythmia
* patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient older than 18 years hospitalized in neuro-intensive care unit with a "non-severe" subarachnoid hemorrhage (WFNS 1 or 2)
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2020-12-25 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Global Longitudinal Strain | Day 1 of hospitalization
  It is calculated using values of longitudinal strain measured in the three-,four-, and two-chamber of the left ventricle of the heart. GLS is expressed as percentage. Strain is a measure of myocardial muscle fiber shortening during contraction and is calculated as the systolic segment shortening between end-systolic (ES) segment length (L) and end-diastolic (ED) length: strain = (-LES - LED)/LED x 100 %.

SECONDARY OUTCOMES:
Global Longitudinal Strain | Day 3 of hospitalization
  is calculated using values of longitudinal strain measured in the three-,four-, and two-chamber of the left ventricle of the heart. GLS is expressed as percentage. Strain is a measure of myocardial muscle fiber shortening during contraction and is calculated as the systolic segment shortening between end-systolic (ES) segment length (L) and end-diastolic (ED) length: strain = (-LES - LED)/LED x 100 %.
Global Longitudinal Strain | Day 7 of hospitalization
  is calculated using values of longitudinal strain measured in the three-,four-, and two-chamber of the left ventricle of the heart. GLS is expressed as percentage. Strain is a measure of myocardial muscle fiber shortening during contraction and is calculated as the systolic segment shortening between end-systolic (ES) segment length (L) and end-diastolic (ED) length: strain = (-LES - LED)/LED x 100 %.
Change of Left Ventricular Ejection Fraction using Simpson technique | Days 1, 3 and 7 of hospitalization
Change in serum troponin level | Days 1, 3 and 7 of hospitalization
Change in brain natriuretic peptide (BNP) level | Days 1, 3 and 7 of hospitalization
Electrocardiogram abnormalities | Up to day 7 of hospitalization
  Abnormalities expected:
  * abnormal Q or QS wave (≥30 ms or a pathological R wave in V1 to V2)
  * ST de- pression (ST depression ≥ 0.1 mV, 80 ms post-J point)
  * ST elevation (ST elevation ≥ .1 mV)
  * peaked upright T wave (prominent peaked T wave)
  * T-wave inver- sion (pathologic T-wave inversion)
  * nonspecific ST- or T-wave changes

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No